CLINICAL TRIAL: NCT06775353
Title: The Effect of Dexamethasone Eye Drops on Retinopathy of Prematurity, a Swedish Registry-based Study
Brief Title: To Assess the Effect of Dexamethasone Eye Drops on the Retinopathy of Prematurity Outcome
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-05824-01
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Retinopathy of Prematurity (ROP)
Keywords: topical dexamethasone
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all screened infants for ROP borne before week 30 in four swedish regions: The treatment frequency for severe ROP was compared between the control years 2015-2018 and the intervention years 2020-2021, but also for all children screened during these years. One region introduced dexamethasone eye drops during the intervention years. The other three regions did not and thus served as a control group.
  Interventions: Drug: Dexamethasone eyedrop

INTERVENTIONS:
Drug: Dexamethasone eyedrop — Infants who developed stages of pretreatment-requiring severe ROP were usually given one eyedrop of dexamethasone daily until the ROP changes regressed.

SUMMARY:
The purpose is to compare the treatment frequency of preterm infants who developed severe Retinopathy of Prematurity (ROP) during the years 2015-2018 with 2020-2021 in the country, using the statistical method 'difference in differences' to investigate the potential for scientific evidence regarding the introduction of dexamethasone eye drops' effect on the development of severe treatment-requiring ROP. During these years, the investigatots assess that the recommended oxygen saturation levels for preterm infants have remained stable at each clinic, which will serve as its own reference.

DETAILED DESCRIPTION:
Retinopathy of Prematurity (ROP) can develop in premature infants and involves abnormal growth of blood vessels in the retina. It can lead to severe visual impairment or blindness if not treated in time. In Sweden, approximately 40-50 children require treatment for severe ROP each year. Children at the highest risk are screened to detect ROP at an early stage, and, if necessary, laser treatment of the retina is performed or an injection of an anti-vascular endothelial growth factor (anti-VEGF) agent is administered. However, laser treatment burns away the outermost part of the retina, and anti-VEGF carries a significant risk of recurring treatment needs, resulting in increased anesthesia and examination sessions for the child, risk of eye infection, lens damage, and uncertainty about the drug's broader effects on the child's brain or body.

Dexamethasone is a corticosteroid commonly used in eye drop form to treat inflammatory and angiogenic eye diseases. Dexamethasone is also administered systemically in neonatal care to treat lung disease and wean premature infants off ventilator support, often in relatively high doses early in the infant's life.

Increased inflammation in the eyes has been reported in ROP. According to both national and several international guidelines, dexamethasone eye drops are administered in tapering doses after laser treatment for severe ROP, often staring with 1 drop 3 times daily. When a child begins developing severe ROP, it is classified as Type-1 ROP and Type-2 ROP. Type-1 ROP requires treatment within 72 hours, while Type-2 ROP is considered a precursor to Type-1 ROP.

In the Southern Healthcare Region of Sweden, the investigators have initiated earlier use of low dose dexamethasone eye drops, specifically when it appears that the child is transitioning from Type-2 ROP to Type-1 ROP. Usually 1 drop daily. In a pilot study published in September 2021, the investigators observed that only 24% of children who received dexamethasone eye drops at Type-2 ROP progressed to Type-1 ROP, compared to 74% of children who did not receive dexamethasone eye drops for the same type of ROP.

In Sweden, there is a national quality registry for ROP care, SWEDROP, with approximately 98% coverage. The investigators now aim to conduct a study based on this quality registry and compare the results from the Southern Healthcare Region with other regions in Sweden that have not used dexamethasone for Type-2 ROP. The goal is to determine whether the "difference-in-differences" method can provide stronger scientific evidence supporting this treatment approach. The plan is to compare the number of children who progressed to laser treatment in the years before the introduction of dexamethasone for Type-2 ROP with data from 2020-2021, when almost all children in the Southern Healthcare Region, received dexamethasone for Type-2 ROP. Specifically, the investigators will compare the years 2015-2018 with 2020-2021. The year 2019 served as a transitional period in the Southern Healthcare Region, where children were treated with varying doses, and therefore it will not be included in the primary comparison. The treatment frequency will be analyzed both for all screened children and specifically for those who developed severe ROP. Severe ROP is defined as type 1 and type 2 ROP.

Age at treatment will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

- During 2015-2018 and 2020-2021, all children born before week 30 in the Southern Health Region and three regions where dexamethasone eye drops were not used to prevent severe treatment-requiring ROP were included

Exclusion Criteria:

If a child has not completed the screening examinations for ROP-

Min Age: 31 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Between 2015-2018 and 2020-2021, all children born before week 30 in the Southern Healthcare Region and three other regions where dexamethasone eye drops were not used to prevent severe treatment-requiring ROP were included in the study population. A specific analysis was conducted on the children who developed severe ROP, Type 1 and Type 2 ROP.
Sampling Method: Non-Probability Sample
Enrollment: 2017 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Show the clinical effect of dexamethasone eyedrops in reducing treatment-requiring severe ROP | The treatment frequency was compared for the intervention group with the control group during the control years 2015-2018 and the intervention years 2020-2021 when dexamethasone eye drops were introduced in the intervention group.
  Has the treatment frequency of severe ROP decreased in the Southern healthcare region compared to other healthcare regions after the introduction of early low-dose corticosteroid treatment in the form of eye drops? Treatment frequency will also be analyzed for all children screened during these years. The statistical method difference in differences will be used in the analyses.
  Age at treatment will also be studied to see if the cortisone drops affect this factor.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Sciences, Ophthalmology, Lund University, Skåne University Hospital, Lund, Sweden, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rivera JC, Holm M, Austeng D, Morken TS, Zhou TE, Beaudry-Richard A, Sierra EM, Dammann O, Chemtob S. Retinopathy of prematurity: inflammation, choroidal degeneration, and novel promising therapeutic strategies. J Neuroinflammation. 2017 Aug 22;14(1):165. doi: 10.1186/s12974-017-0943-1. PMID 28830469
- [Background] Doyle LW, Cheong JL, Ehrenkranz RA, Halliday HL. Early (< 8 days) systemic postnatal corticosteroids for prevention of bronchopulmonary dysplasia in preterm infants. Cochrane Database Syst Rev. 2017 Oct 24;10(10):CD001146. doi: 10.1002/14651858.CD001146.pub5. PMID 29063585
- [Background] Chiang MF, Quinn GE, Fielder AR, Ostmo SR, Paul Chan RV, Berrocal A, Binenbaum G, Blair M, Peter Campbell J, Capone A Jr, Chen Y, Dai S, Ells A, Fleck BW, Good WV, Elizabeth Hartnett M, Holmstrom G, Kusaka S, Kychenthal A, Lepore D, Lorenz B, Martinez-Castellanos MA, Ozdek S, Ademola-Popoola D, Reynolds JD, Shah PK, Shapiro M, Stahl A, Toth C, Vinekar A, Visser L, Wallace DK, Wu WC, Zhao P, Zin A. International Classification of Retinopathy of Prematurity, Third Edition. Ophthalmology. 2021 Oct;128(10):e51-e68. doi: 10.1016/j.ophtha.2021.05.031. Epub 2021 Jul 8. PMID 34247850
- [Background] Holmstrom G, Hellstrom A, Granse L, Saric M, Sunnqvist B, Wallin A, Tornqvist K, Larsson E. New modifications of Swedish ROP guidelines based on 10-year data from the SWEDROP register. Br J Ophthalmol. 2020 Jul;104(7):943-949. doi: 10.1136/bjophthalmol-2019-314874. Epub 2019 Nov 1. PMID 31676594
- [Background] Ohnell HM, Andreasson S, Granse L. Dexamethasone Eye Drops for the Treatment of Retinopathy of Prematurity. Ophthalmol Retina. 2022 Feb;6(2):181-182. doi: 10.1016/j.oret.2021.09.002. Epub 2021 Sep 10. No abstract available. PMID 34517147